CLINICAL TRIAL: NCT03240120
Title: A Prospective Study of Dabigatran Etexilate as Primary Treatment of Malignancy Associated Venous Thromboembolism
Brief Title: A Study of Dabigatran Etexilate as Primary Treatment of Malignancy Associated Venous Thromboembolism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Eric W.C. Tse, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKU-OTI-01
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Dabigatran; Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabigatran etexilate & Tinzaparin (Experimental): Tinzaparin 175 iu/kg daily will be started after the diagnosis of VTE is confirmed dabigatran 150mg twice daily from Day 6 onward till 6 months after underlying disease remission.
  Interventions: Drug: Dabigatran etexilate; Drug: Tinzaparin

INTERVENTIONS:
Drug: Dabigatran etexilate — Pradaxa 150 mg hard capsules
  Other Names: Pradaxa
Drug: Tinzaparin — Tinzaparin 175 iu/kg daily will be started after the diagnosis of VTE is confirmed

SUMMARY:
This trial aims at determining if dabigatran is effective in the treatment of malignancy associated VTE. Tolerance and safety of dabigatran will also be assessed.

This is a single armed trial of dabigatran in patients with malignancy associated VTE.

The target recruitment is 99 consecutive patients with active malignancy and newly diagnosed VTE (deep vein thrombosis and/or pulmonary embolism) in Queen Mary Hospital.

Tinzaparin 175 iu/kg daily will be started after the diagnosis of VTE is confirmed (duplex Doppler ultrasonography for deep vein thrombosis, and computed tomography for pulmonary embolism), and a written consent is obtained. Patients will be switched to dabigatran 150mg twice daily from day 6 onwards. The first dose of dabigatran will be given within 2 hours before the time that the next dose of tinzaparin would have been due. Anticoagulation will be continued as long as malignancy is active. If patients achieve a complete remission of their underlying malignancies, dabigatran will be continued for 6 months further.

DETAILED DESCRIPTION:
Patients with malignancies are at increased risks of venous thromboembolism (VTE). The annual incidence of VTE in cancer patients is 0.5%, which is 5-fold more than the general population . Low molecular weight heparin (LMWH) has been the standard treatment for malignancy-associated VTE. This recommendation follows the results of the Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent VenousThromboembolism in Patients with Cancer (CLOT) trial, which showed superiority of Low molecular weight heparin (LMWH) over warfarin in cancer patients with VTE .

Low molecular weight heparin (LMWH) has a number of inherent advantages over warfarin. It does not interact with chemotherapeutic agents, and dose titration is not necessary. Furthermore, the risks of both bleeding and breakthrough VTE are also lower with LMWH. However, the requirement of daily subcutaneous injection makes LWMH inconvenient to use. Most patients have difficulties continuing daily injection, partly owing to compliance issues, but also because an emaciated state in some patients makes subcutaneous injection painful. As the life expectancy of solid cancer patients is improved with novel treatment options, the choice of anticoagulation has become a major issue in the management of VTE in this patient population.

The main reason underlying the inferior performance of warfarin in oncology patients is difficult dose titration. Drug interaction and hepatic dysfunction are common in patients on chemotherapy. Frequent interruptions of warfarin for invasive procedures and chemotherapy-induced-thrombocytopenia also lead to fluctuations in anticoagulation level. As a result, highs risk of recurrence of VTE and bleeding were observed in cancer patients taking warfarin. Direct-acting oral anticoagulants (DOACs), on the other hand, may be an attractive alternative treatment to LMWH. They are administered at a fixed dose with predictable pharmacokinetics, so that therapeutic monitoring is not required. There is minimal food and drug interaction. They have been shown to be effective in the treatment of VTE in several pivotal randomized controlled trials in comparison with warfarin . However, their role in malignancy associated VTE is yet to be determined, because cancer patients were either excluded or very much underrepresented in these VTE treatment trials. Moreover, the non-inferiority of DOACs in VTE treatment was only demonstrated against warfarin, which is already shown to be suboptimal in oncology patients. A trial directly comparing DOACs with LMWH in malignancy associated VTE is therefore needed.

Dabigatran etexilate is an oral thrombin inhibitor. It was shown in the RECOVER study to be effective in treatment of VTE and it has a lower bleeding risk than warfarin. It is not metabolized by cytochrome P450 system and therefore, in contrast to other DOACs, concomitant administration of CYP3A4 inducers or inhibitors is not a concern.

We propose this prospective single armed trial to evaluate the efficacy and safety of dabigatran in the treatment of malignancy associated VTE. We will compare the result with our historical control who were treated with LMWH.

ELIGIBILITY:
Inclusion Criteria:

1. are aged 18 years or above;
2. have acute symptomatic deep vein thrombosis or pulmonary embolism with objective confirmation;
3. have active cancer, which is defined as a diagnosis of cancer other than basal cell or squamous cell carcinoma of skin within six months before enrollment, any treatment for cancer within the previous six months or recurrent or metastatic cancer.
4. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
5. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. have Eastern Cooperative Oncology Group (ECOG) performance status score of > 2 at the time of randomization;
2. have life expectancy of less than 3 months;
3. have active bleeding, are at high risk of bleeding, or have contraindications to anticoagulant treatment;
4. receive thrombectomy or fibrinolytic agent to treat the current episode of VTE;
5. receive more than 72 hours pre-treatment with therapeutic dosages of anticoagulant treatment prior to randomization to treat the current VTE episode;
6. are already on long term oral anticoagulation;
7. are on low molecular weight heparin for indications other than VTE;
8. have platelet count of less than 100 x 109/L;
9. are on dual antiplatelet therapy;
10. have a serum creatinine level of more than 220 umol/L or have a calculated creatinine clearance (CrCl) of less than 30 ml/min;
11. have alanine aminotransferase level more than 2 times the upper limit of normal range or cirrhosis;
12. have history of heparin induced thrombocytopenia;
13. are on treatment of potent inhibitors or inducers of P-glycoprotein.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with symptomatic VTE | up to 2 years
  first episode of objectively documented symptomatic recurrent VTE (deep vein thrombosis, pulmonary embolism)

SECONDARY OUTCOMES:
number of mortality, clinically relevant major and non-major bleeding | up to 2 years
  bleeding (major and non-major) and death

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Hwang, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided